CLINICAL TRIAL: NCT00851812
Title: Aerobic and Resistance Exercise for Cancer Treatment-Related Fatigue
Brief Title: Exercise for Breast Cancer Patients (EXCAP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Karen Mustian, Associate Professor, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 8029NCI
Record Dates: First submitted 2009-02-24; First posted 2009-02-26 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Fatigue
Keywords: Exercise; Breast cancer; fatigue
MeSH Terms: conditions — Fatigue; Motor Activity; Breast Neoplasms | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Other): Usual Care: Standard care monitoring
  Interventions: Behavioral: Exercise
- Arm 2 (Experimental): Progressive walking and resistance exercise treatment
  Interventions: Behavioral: Progressive walking and resistance exercise treatment

INTERVENTIONS:
Behavioral: Exercise — Standard care monitoring
  Other Names: Usual care: standard care monitoring
  Arms: Arm 1
Behavioral: Progressive walking and resistance exercise treatment — Home-based exercise : Progressive walking and resistance program
  Arms: Arm 2

SUMMARY:
The purpose of this study is to examine if exercise helps improve cancer-related fatigue.

Hypothesis: A structured home-based walking and progressive resistance exercise program will be efficacious in relieving cancer-related fatigue, preventing aerobic and anaerobic deconditioning and skeletal muscle wasting, as well as improving inflammatory cytokine profiles in breast cancer survivors as well as those receiving radiation treatment.

DETAILED DESCRIPTION:
Fatigue is a frequently reported side effect of cancer treatment. Fatigue related to cancer and its treatment is different from fatigue occurring in other situations and its specific causes have not been identified. Exercise may or may not improve this type of fatigue. The purpose of this study is to examine how cancer treatments impact normal lifestyle physical activity patterns and participation in physical activity, as well as the ability of a walking and progressive resistance exercise program to reduce cancer-related fatigue in breast cancer patients. This study also examines if the walking and progressive resistance exercise program improves other factors such as quality of life, depression, anxiety, ability to sleep, self esteem, cardiovascular fitness, energy expenditure, muscular strength, muscle mass, and immune function (as measured by inflammatory cytokines).

ELIGIBILITY:
Inclusion Criteria:

* Have a primary diagnosis of breast cancer,
* Have a functional capacity rating of 60 or greater on the Karnofsky Performance Scale, when assessed by the oncologist (or physician's designee)
* Be breast cancer survivor(e.g., surgery, radiation therapy, chemotherapy, hormone therapy). Have a life expectancy of >1 year as determined by the patient's oncologist.
* Have the approval of their treating physician, study physician(or physician's designee) to participate in sub-maximal physiological fitness testing and a low to moderate home-based walking and progressive resistance exercise program.
* Be able to read English.
* Be 21 years of age or older.
* Give informed consent.

Exclusion Criteria:

* Have bone metastases that preclude participation in an exercise program either due to symptoms such as pain or location of bone metastasis.
* Have physical limitations (i.e. cardiorespiratory, orthopedic, central nervous system) that contraindicate participation in sub-maximal physiological fitness testing, or a low to moderate home-based walking and progressive resistance program, as assessed by the PAR-Q and radiation oncologist (or physician's designee)
* Be identified as in the Active or Maintenance Stage of exercise behavior as assessed by the 1-item Exercise Stages of Change Short Form.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2007-05; Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Cancer-related fatigue | 4.5 months

SECONDARY OUTCOMES:
To provide preliminary data on influence of QOL and it's relationship to CRF | 4.5 months

CONTACTS AND LOCATIONS:
Overall Officials: Karen Mustian, Ph.D., Principal Investigator — James P. Wilmot Cancer Center, University of Rochester
Locations (1):
- James P. Wilmot Cancer Center, University of Rochester, Rochester, New York, United States